CLINICAL TRIAL: NCT01521078
Title: Randomized Controlled Trial of a Brief Personalized Feedback Intervention in University Students
Brief Title: Web-based Personalized Feedback for University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: University of Houston (Other)
Responsible Party: Principal Investigator, John Cunningham, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CAMH#152/2011
Record Dates: First submitted 2012-01-26; First posted 2012-01-30 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-05

CONDITIONS: Risky Alcohol Consumption

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Provided access to the Check Your Drinking University version (CYDU).
  Interventions: Behavioral: Check Your Drinking University version
- Control (No Intervention): No invention control group

INTERVENTIONS:
Behavioral: Check Your Drinking University version — The CYDU is an internet-based intervention that provides a personalized feedback summary which compares the participant's drinking to that of other university students. The CYDU is a modified version of the Check Your Drinking screener which has been validated in four separate randomized controlled trials. The primary modification of the CYDU is that the population norms used for comparison are those of university students (in the USA or Canada).
  Arms: Intervention

SUMMARY:
Excessive alcohol consumption in university students continues for be a serious public health concern with a variety of negative consequences. There have been a number of different brief interventions developed to address this issue among university students. The current project will add to this literature by evaluating the use of a personalized feedback intervention (www.CheckYourDrinkingU.net; CYDU). Specifically, this trial will examine whether providing access to the CYDU will result in short-term reductions in drinking. This issue is important as use of these interventions is not a mandatory requirement for university students so the issue is whether making materials of this type available leads to any reductions in risky drinking. It is hypothesized that students provided access to the CYDU will display greater reductions in drinking at a six-week follow-up as compared to students who were not provided access to the CYDU.

ELIGIBILITY:
Inclusion Criteria:

* AUDIT-C score of 4 or more at baseline

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 425 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Alcohol Use Disorders Identification Test - Consumption scale (AUDIT-C scale) | 6 weeks
  AUDIT-C is a scale that is a composite of three items - frequency of alcohol use, drinks per drinking day, and frequency of 5+ drinking occasions. Scores ranges from 0 to 12 with higher scores indicating more severe alcohol problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Cunningham JA, Neighbors C, Bertholet N, Hendershot CS. Use of mobile devices to answer online surveys: implications for research. BMC Res Notes. 2013 Jul 8;6:258. doi: 10.1186/1756-0500-6-258. PMID 23834999
- [Derived] Cunningham JA, Hendershot CS, Murphy M, Neighbors C. Pragmatic randomized controlled trial of providing access to a brief personalized alcohol feedback intervention in university students. Addict Sci Clin Pract. 2012 Oct 10;7(1):21. doi: 10.1186/1940-0640-7-21. PMID 23185985